CLINICAL TRIAL: NCT01410175
Title: "Impact on the Incidence of Surgical Site Infection in Abdominal Gynecological Surgery by Comparing the Skin and Subcutaneous Tissue Incision With Cold Scalpel and Electrocautery in a Period of Two Years."
Brief Title: Comparison of the Impact of Electric Scalpels Versus Cold Scalpels
Acronym: SCL01
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Barretos Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SCALPEL 01
Record Dates: First submitted 2011-06-21; First posted 2011-08-04 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Wound Infection; Cicatrization
MeSH Terms: conditions — Wound Infection; Cicatrix

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional scalpel (Experimental): Use of conventional scalpel to incise the skin and subcutaneous layer.
  Interventions: Device: Conventional scalpel
- Electric scalpel (No Intervention): Use of electric scalpel to incise the skin and subcutaneous layer.

INTERVENTIONS:
Device: Conventional scalpel — Use of conventional scalpel to incise the skin and subcutaneous layers.
  Other Names: Cold scalpel
  Arms: Conventional scalpel

SUMMARY:
Surgical site infection (SSI) is the second commonest hospital infection, despite advances in prevention that have been achieved.

According to Fernàndes, experimental studies have demonstrated that incorrect use of electric scalpels may double the rate of SSI during electrocauterization.

Because of the lack of solid data in the literature, in relation to the impact on SSI of using electric scalpels for making incisions in the skin and all subcutaneous tissues, it was judged to be opportune to conduct the present study.

Objectives:

* To compare the incidence of SSI and other complications of the operative wound among patients undergoing elective abdominal gynecological surgery at Barretos Cancer Hospital, between the use of electric and cold scalpels.
* To identify the incidence of SSI and other complications of the operative wound among patients undergoing elective abdominal gynecological surgery, when using electric scalpels for skin incisions and for subcutaneous incisions.
* To identify the main risk factors for SSI among patients undergoing elective abdominal gynecological surgery.

DETAILED DESCRIPTION:
Introduction Surgical site infection (SSI) is the second commonest hospital infection, despite advances in prevention that have been achieved. However, among surgical patients, it is the hospital infection of greatest incidence. In the United States, it has been estimated that around 500,000 cases of SSI occur every year, thus generating an annual cost of more than 1.6 billion dollars.

According to the Centers for Disease Control (CDC), SSI can appear up to 30 days after performing the surgical procedure and up to one year afterwards, when a prosthesis was implanted. SSI is classified as superficial infection when it only affects the skin and subcutaneous tissue at the incision site. It is classified as deep infection when it involves deep structures of the wall and muscle layers of organs and spaces in any part of the anatomy that is opened or manipulated during the surgical procedure, with the exception of the incision.

SSI has a series of consequences. These include increased duration of hospitalization, increased cost of medical and hospital care, increased prescription of broad-spectrum antibiotics (with consequent increased bacterial resistance) and increased postoperative mortality, given that 30% to 40% of deaths during this period result from this type of infection.

The risk factors most frequently correlated with SSI are in connection with the patient and the surgical procedure and include obesity, malnutrition, smoking, age extremes, diabetes, chronic obstructive pulmonary disease, immunosuppression, alcoholism, use of corticoids, potential for contamination of the operative wound, long-duration operations, presence of a foreign body at the surgical site, incorrect administration of antibiotic prophylaxis and poor surgical technique. Thus, the risk of SSI may vary according to the type of surgery and each individual's inherent conditions.

With regard to surgical technique, the points that need to be taken into consideration include careful dissection and manipulation of the tissue so as to minimize the tissue trauma, adequacy of hemostasis to impede formation of hematomas, avoidance of environments favorable to microbe proliferation and excessive use of electric scalpels or their use with higher-than recommended currents, which has a high potential for tissue devitalization. According to Fernàndes, experimental studies have demonstrated that incorrect use of electric scalpels may double the rate of SSI during electrocauterization.

Because of the lack of solid data in the literature, in relation to the impact on SSI of using electric scalpels for making incisions in the skin and all subcutaneous tissues, it was judged to be opportune to conduct the present study.

Objectives:

* To compare the incidence of SSI and other complications of the operative wound among patients undergoing elective abdominal gynecological surgery at Barretos Cancer Hospital, between the use of electric and cold scalpels.
* To identify the incidence of SSI and other complications of the operative wound among patients undergoing elective abdominal gynecological surgery, when using electric scalpels for skin incisions and for subcutaneous incisions.
* To identify the main risk factors for SSI among patients undergoing elective abdominal gynecological surgery.

Methodology:

This is a blinded randomized clinical trial composed of two groups (cold scalpel versus electric scalpel), among patients undergoing elective abdominal gynecological surgery at Barretos Cancer Hospital between July 2010 and July 2012. These patients will fulfill the following inclusion criteria: over 18 years of age, agreement to participate in the study and undergoing elective abdominal gynecological surgery for the purposes of diagnosis or curative or palliative oncological treatment. The following types of patient will be excluded: patients undergoing surgery with manipulation of the digestive system, patients undergoing surgery to open a stoma and cases of reoperation. The randomization will be performed at the time of the surgery by the Research Support Center of Barretos Cancer Hospital, with further subdivision of the patients into two groups, with body mass index (BMI) < 30 and ≥ 30. The cold scalpel and electric scalpel will be used in accordance with the randomization, to open the skin and the subcutaneous cellular tissue. The aponeurosis and peritoneum will be incised using an electric scalpel. The data will be gathered by the investigator, who will make direct observations of the operative wound in order to make diagnoses of SSI after discharge from hospital, with assessments on the 14th and 30th days after the operation. The present project has been approved by the Research Ethics Committee of Barretos Cancer Hospital. Subjects who agree to participate will show their acceptance through signing a free and informed consent statement. Other factors such as hematoma, seroma, bulging, etc., will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* age => 18 yo
* elective abdominal gynecological surgery for the purposes of diagnosis or curative or palliative oncological treatment

Exclusion Criteria:

* surgery with manipulation of the digestive system
* cases of re-operation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2010-07; Primary Completion 2012-07 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change in Surgical Incision Complications | 15 and 30 days after surgery
  The following complications will be analyzed in those days: site infection, seroma, dehiscence, hematoma, bruise, hyperemia and quality of healing.

CONTACTS AND LOCATIONS:
Overall Officials: Regiane L Rongetti, Principal Investigator — Barretos Cancer Hospital
Locations (1):
- Barretos Cancer Hospital, Barretos, São Paulo, Brazil

REFERENCES:
- [Derived] Rongetti RL, Oliveira e Castro Pde T, Vieira RA, Serrano SV, Mengatto MF, Fregnani JH. Surgical site infection: an observer-blind, randomized trial comparing electrocautery and conventional scalpel. Int J Surg. 2014;12(7):681-7. doi: 10.1016/j.ijsu.2014.05.064. Epub 2014 May 24. PMID 24866067